CLINICAL TRIAL: NCT02915991
Title: Prospective, Single Arm, Open Label, User Evaluation Sudy of SyncVision System With Software v4.X
Brief Title: User Evaluation Study of SyncVision System With Software v4.X
Acronym: Prepare II
Status: Terminated | Type: Observational
Why Stopped: slow recruitment and change in regulatory landscape
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-CV-001
Record Dates: First submitted 2016-06-16; First posted 2016-09-27 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary catheterization; Instantaneous wave free ratio (iFR); Fractional Flow Reserve (FFR); automated co-registration
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: This is a single-arm study, so all patients enrolled will be in this arm and will undergo diagnostic catheterization procedure as per standard hospital care.

SUMMARY:
This is a prospective, single-arm, unblinded, case observation study evaluating a commercially released 'Conformité Européenne' (CE)-mark co-registration software system along-side of a commercially- released CE-mark coronary physiology and X-ray system during routine clinical workflow. The purpose of this study is to collect Professional user feedback regarding clinical utility of the SyncVision 4.X system.

DETAILED DESCRIPTION:
The PREPARE II study will enroll a maximum of 200 patients in up to 5 sites. No follow-up will be performed. The PREPARE II study will only collect data during diagnostic angiogram or percutaneous coronary intervention (PCI) procedure, when performed as per standard hospital care.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible and indicated for cardiac catheterization and pressure-wire assessment in the coronary arteries as per standard hospital practice
* Males over the age of 18 years and post-menopausal females
* Patient is able to give written informed consent prior to using his/her study data for evaluation and documentation

Exclusion Criteria:

- Patient is unable to give written informed consent prior to using his/her study data for evaluation and documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiets that undergo a cardiac catheterization and pressure-wire assessment in the coronary arteries as per standard hospital practice.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Professional user feedback regarding clinical utility of the SyncVision 4.X system | Day 1 (Post-Procedure)
  After the procedure the physician will be asked to rate and comment on the clinical utility and features of the SyncVision 4.X system in the post-study user evaluation questionnaire. This will include questions on the potential of the system to facilitate clinical decision-making, utility of co-registration workflow and functionality, quality of the co-registration and user interface functions.

SECONDARY OUTCOMES:
Difference between assessments | Day 1 (Post-Procedure)
  Differences between the clinical assessment based on the existing time-based pullback graph and clinical assessment based on the automated co-registration of pullback graph with the angio image are performed by using a rating system 1 - 5 (1=Unacceptable, …., 5=Excellent).
  The co-registration and functionality points assessed are:
  * Workflow associated with achieving Physiology values co-registration
  * Physiology values co-registration results display clear and functionality convenient for use
  * Angiogram & Roadmap selection
  * Auto roadmap generation
  * Pathway indication and correction
  * Co-Registration sequence: Roadmap-navigation and calibrated graph navigation
  * Length measurements
Distinguish tandem, diffuse and mixed disease | Day 1 (Post-Procedure)
  Ability to distinguish tandem, diffuse and mixed disease based on the physiological pullback profile display and the co-registered physiological pullback profile display are performed by the use of a rating system 1 - 5 (1=Unacceptable, …., 5=Excellent). The points assessed and compared are:
  * Distinguish tandem lesions
  * Distinguish diffuse diseased lesions
  * Distinguish mixed diseased lesions
Comparison of pre-intervention expected distal-most iFR with post-intervention actual distal-most iFR values | Day 1 (Post-Procedure)
  Comparison of the pre-intervention expected distal-most iFR with the post-intervention actual distal-most iFR values is based on the comparison of real time pre- and post-intervention displayed iFR values on the physiological pullback profile display and the co-registered physiological pullback profile display.The points assessed and compared are:
  * Pre-intervention distal most iFR
  * Post-intervention iFR

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Frimerman, Professor, Principal Investigator — The medical research and development fund for health services Hillel Yafe; Ariel Roguin, Professor, Principal Investigator — Rambam Healthcare Campus
Locations (2):
- Israel (2):
  - The medical research and development fund for health services Hillel Yaffe, Hadera
  - Rambam Health Corporation, Haifa

IPD SHARING:
Plan to Share IPD: No